CLINICAL TRIAL: NCT03538314
Title: A Phase I, Open-label, Multicenter Study Investigating the Tolerability and Efficacy of UV1 Vaccine in First-line Malignant Melanoma Patients Planned for Treatment With Pembrolizumab
Brief Title: UV1 Vaccine With Pembrolizumab for Patients With Unresectable or Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ultimovacs ASA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UV1/hTERT-MM-103
Record Dates: First submitted 2018-04-22; First posted 2018-05-29 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: UV1/GM-CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Treatment (Experimental): UV1/GM-CSF
  Interventions: Drug: UV1; Drug: GM-CSF

INTERVENTIONS:
Drug: UV1 — UV1 (300 microgram)
Drug: GM-CSF — GM-CSF (37,5 or 75 microgram)

SUMMARY:
UV1 is a therapeutic cancer vaccine that has been explored in prostate and lung cancers, and in combination with ipilimumab in malignant melanoma. This study will explore the safety, tolerability and efficacy of UV1 administered with GM-CSF in melanoma patients who are also receiving pembrolizumab.

ELIGIBILITY:
Key Inclusion Criteria:

1. Stage IIIB, IIIC or IV melanoma
2. Previously untreated and eligible for pembrolizumab treatment (prior treatment with BRAF and MEK inhibitors permitted) 3) Adequate blood, liver and kidney function 4) Consent to undergo tumor biopsies during the study

Exclusion Criteria:

1. Uveal or ocular malignant melanoma
2. History of hematologic or primary solid tumor malignancy with the exception of patients in remission for at least 5 years, as judged by the investigator are allowed
3. Prior systemic treatment for unresectable or metastatic melanoma. Exception: Prior treatment with BRAF and MEK inhibitors permitted. A washout period of at least 3-half-lives (median terminal half-life) prior to the first dose of trial treatment must have elapsed.
4. Prior therapy with an anti-CTLA4, anti-PD-1, anti-PD-L1, anti-PD-L2 agent or oncolytic virus.
5. Known hypersensitivity to GM-CSF
6. Women who are breastfeeding, pregnant or expect to be pregnant during the study through 6 months after the last dose
7. Men who plan to become a father during the study through 4 months after the last dose of study medication
8. Known history of, or any evidence of active, non-infectious pneumonitis
9. History of cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment-related adverse events | Up to week 29
  Frequency and severity of adverse events

SECONDARY OUTCOMES:
Tumor response | Up to week 52
  RECIST and iRECIST
The length of time from the start of treatment that patients are still alive. | up to 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - John Wayne Cancer Center, Santa Monica, California
  - University of Iowa Carver College of Medicine, Iowa City, Iowa
  - St. Luke's University Health Network, Easton, Pennsylvania
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah